CLINICAL TRIAL: NCT07346235
Title: OPTIMAL-DOSE: A Randomized, Open-Label, Non-Inferiority Trial Comparing Fixed Daily Doses of 150 IU Versus 225 IU of Follicle-Stimulating Hormone in Predicted Normal Responders Undergoing In Vitro Fertilization/Intracytoplasmic Sperm Injection
Brief Title: 150 IU vs. 225 IU FSH in Normal Responders: The OPTIMAL-DOSE Trial
Acronym: OPTIMAL-DOSE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: American Hospital 2 Kosovo (Other)
Responsible Party: Principal Investigator, Goksu Goc, Principal Investigator, American Hospital 2 Kosovo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMAL-DOSE-2026-001
Record Dates: First submitted 2025-12-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female
Keywords: IVF; ICSI; FSH; Gonadotropin; Ovarian Stimulation; Normal Responder; Live Birth Rate; OHSS
MeSH Terms: conditions — Infertility, Female | interventions — Follicle Stimulating Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 150 IU FSH Group (Experimental): Participants receive a fixed daily dose of 150 IU of recombinant or urinary FSH starting on day 2-3 of the menstrual cycle, continuing until trigger day.
  Interventions: Drug: Follicle-stimulating hormone (FSH)
- 225 IU FSH Group (Active Comparator): Participants receive a fixed daily dose of 225 IU of recombinant or urinary FSH starting on day 2-3 of the menstrual cycle, continuing until trigger day.
  Interventions: Drug: Follicle-stimulating hormone (FSH)

INTERVENTIONS:
Drug: Follicle-stimulating hormone (FSH) — Daily subcutaneous injection of 150 IU FSH
  Arms: 150 IU FSH Group
Drug: Follicle-stimulating hormone (FSH) — Daily subcutaneous injection of 225 IU FSH
  Arms: 225 IU FSH Group

SUMMARY:
This is a single-center, randomized, open-label, non-inferiority trial comparing two fixed daily doses of follicle-stimulating hormone (FSH): 150 IU versus 225 IU in women with predicted normal ovarian response undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) with a gonadotropin releasing hormone (GnRH) antagonist protocol. The primary objective is to determine whether the 150 IU dose is noninferior to the 225 IU dose regarding the cumulative live birth rate per initiated cycle. Secondary objectives include comparing oocyte yield, incidence of OHSS, treatment costs, and patient-reported outcomes.

DETAILED DESCRIPTION:
Background: Controlled ovarian stimulation (COS) with exogenous FSH is a cornerstone of IVF treatment. The optimal starting dose of FSH for women with normal ovarian reserve remains controversial, with doses ranging from 150 IU to 300 IU used in clinical practice.

Both 150 IU and 225 IU are widely used, but no randomized controlled trial has directly compared these two specific doses in predicted normal responders.

Objective: To determine if a fixed daily dose of 150 IU FSH is non-inferior to 225 IU FSH with respect to cumulative live birth rate per initiated cycle.

Methods: A total of 440 women (220 per group) will be randomized 1:1 to receive either 150 IU or 225 IU of FSH daily, starting on day 2-3 of the menstrual cycle. All participants will follow a standard GnRH antagonist protocol. The primary outcome is cumulative live birth rate, defined as the delivery of at least one live-born infant at ≥24 weeks of gestation from the first fresh or any subsequent frozen embryo transfer from a single stimulation cycle. The non-inferiority margin is set at -10% (absolute difference).

Significance: If 150 IU is proven non-inferior, this would support the use of a lower dose, potentially reducing treatment costs and the risk of ovarian hyperstimulation syndrome (OHSS) without compromising efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) 18-30 kg/m².
2. Predicted normal ovarian reserve:
3. Anti-Müllerian Hormone (AMH) 1.2-3.5 ng/mL (measured within 12 months), AND Antral Follicle Count (AFC) 8-20 (both ovaries combined, measured on day 2-5 of the cycle).
4. First or second IVF/ICSI cycle.
5. Planned GnRH antagonist protocol.
6. Both ovaries present and accessible.
7. Written informed consent provided voluntarily.

Exclusion Criteria:

1. Predicted poor or high ovarian response (AMH <1.2 or >3.5 ng/mL; AFC <8 or >20).
2. Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria.
3. Severe endometriosis (Stage III-IV per ASRM).
4. Severe uterine abnormalities affecting implantation.
5. Previous complete fertilization failure (fertilization rate <30%).
6. Severe male factor (sperm count <5 million/mL, or requirement for donor sperm/TESE).
7. Uncontrolled endocrine disorders (uncontrolled hypothyroidism, hyperprolactinemia, diabetes).
8. Contraindications to pregnancy or gonadotropins.
9. Participation in another clinical trial within 30 days.
10. Inability to provide informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Cumulative Live Birth Rate per Initiated Cycle | Up to 12 months after randomization
  The delivery of at least one live-born infant at ≥24 weeks of gestation resulting from the first fresh embryo transfer or any subsequent frozen embryo transfer from a single stimulation cycle.

SECONDARY OUTCOMES:
Number of Oocytes Retrieved | Up to 2 weeks
  Total number of oocytes retrieved at oocyte pick-up.
Incidence of Moderate/Severe OHSS | Up to 4 weeks after oocyte retrieval
  Proportion of participants developing moderate or severe OHSS according to Golan classification.
Total FSH Consumption | Up to 2 weeks
  Total amount of FSH (in IU) used during the stimulation cycle.
Clinical Pregnancy Rate | 7 weeks of gestation
  Presence of a gestational sac with fetal heartbeat on ultrasound at 7 weeks of gestation.
Live Birth Rate per Transfer | Up to 12 months after randomization
  Delivery of a live-born infant per embryo transfer procedure.
Cycle Cancellation Rate | Up to 2 weeks
  Proportion of cycles cancelled before oocyte retrieval.

CONTACTS AND LOCATIONS:
Locations (1):
- American Hospital Kosova, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Tilborg TC, Torrance HL, Oudshoorn SC, Eijkemans MJC, Koks CAM, Verhoeve HR, Nap AW, Scheffer GJ, Manger AP, Schoot BC, Sluijmer AV, Verhoeff A, Groen H, Laven JSE, Mol BWJ, Broekmans FJM; OPTIMIST study group. Individualized versus standard FSH dosing in women starting IVF/ICSI: an RCT. Part 1: The predicted poor responder. Hum Reprod. 2017 Dec 1;32(12):2496-2505. doi: 10.1093/humrep/dex318. PMID 29121326